CLINICAL TRIAL: NCT06045416
Title: Extensive Investigation of Immune Responses Against Borrelia Burgdorferi to Improve Diagnosis of Lyme Disease in Children: an Observational Study (BRILLIANT Study)
Brief Title: Borrelia B-cell Diagnostics
Acronym: BRILLIANT
Status: Recruiting | Type: Observational
Sponsor: University Children's Hospital, Zurich (Other)
Collaborators: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-00528
Record Dates: First submitted 2023-09-13; First posted 2023-09-21 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Lyme Disease; Borrelia Infections
Keywords: Borrelia burgdorferi; Lyme disease; Borrelia specific ASCs; Borrelia strains
MeSH Terms: conditions — Lyme Disease; Borrelia Infections | interventions — Spinal Puncture; Arthrocentesis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples With DNA — Blood, serum and blood separated into plasma and peripheral blood mononuclear cells (PBMCs) (DNA) Cerebrospinal fluid (CSF), separated into CSF and CSF-isolated cells (DNA) Synovial fluid (SF), separated into SF and SF-isolated cells (DNA)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- LD_Diff_Diag: LD differential diagnosis cohort: Patients presenting at the ED with differential diagnosis of LD according to the treating physician
  Interventions: Procedure: venous blood puncture
- Heathy_Control: Previously healthy patients (HC) with routine blood investigations presenting at the ED or PID outpatient department
  Interventions: Procedure: venous blood puncture

INTERVENTIONS:
Procedure: venous blood puncture — Venous blood puncture performed at first hospital contact, and at 28 days, 3 month, and 6 months after hospital admission.
  Lumbar puncture and joint puncture for the study will be performed if it is indicated due to diagnostic or therapeutic reasons.
  Other Names: lumbar puncture; joint puncture

SUMMARY:
The investigators propose a single center, prospective observational study in children with Lyme disease (LD), the Borrelia B-cell diagnostics (BRILLIANT) study, to assess the immune response against Borrelia burgdorferi (Bb) with the following main objectives:

1. Development of Bb-specific ASC ELISpot as a new test method for diagnosis of early LD.

   There is an urgent unmet clinical need for a better diagnostic tool for early LD, as the current standard two-tier testing has low sensitivity in recently infected patients and may show false positive results in recovered patients due to long-term persistence of antibodies against Bb. The measurement of Bb-specific ASC with the ELISpot assay my has the potential to overcome these issues and to improve diagnosis in early LD.
2. Extensive analysis of the immune response in LD. The immune response in LD is not well understood. Large-scale studies assessing the detailed immune cell subsets/phenotypes present in blood, CSF, or synovial fluid of LD patients with respective manifestations are lacking.
3. Isolation and characterization of causative Bb species. Existing literature suggests that Bb genospecies and/or genotypes may determine virulence and manifestations, but large-scale studies assessing Bb genospecies/genotypes in different manifestation of LD are lacking.
4. Collection of clinical data about symptoms, severity, routine laboratory and diagnostic test results, treatment, and outcome of LD.
5. Biobanking samples for analysis in the future.

Project population

Inclusion criteria: Children, 0-17 years of age, at University Children's Hospital Zurich:

* LD differential diagnosis cohort: Patients presenting at the ED with differential diagnosis of LD according to the treating physician.
* Control cohort: Previously healthy patients (HC) with routine blood investigations presenting at the ED or PID outpatient department

Exclusion criteria: Primary or secondary immunodeficiency.

DETAILED DESCRIPTION:
Background:

Lyme disease (LD) is the most common tick born disease in Europe. It is caused by an infection with several genospecies of the spirochaetal bacteria Borrelia burgdorferi (Bb).

Although classical disease manifestations are well-known, the clinical presentation in children is often variable and inconclusive, which results in delayed diagnosis and treatment.

Methods/design:

The investigators are conducting an observational cohort study in children with LD. Study site is the University Children's Hospital Zurich. 502 patients will be enrolled. Children from 0-17 years of age presenting with signs and symptoms suspicious for LD are included in the study. Previously healthy children with routine blood investigation are enrolled as healthy controls. Patients will be excluded in cases of primary or secondary immunodeficiency.

Clinical and routine laboratory data regarding course and outcome, as well as venous blood samples are collected at first hospital contact and follow up visits (FUP). FUPs are scheduled at 28 days, 3 months and 6 months after hospital admission. Cerebrospinal fluid (CSF) and synovial fluid (SF) will be collected for the study only if sampling is indicated due to diagnostic or therapeutic reasons.

Primary objectives are to assess Bb-specific ASCs in blood using ELISpot assay, in order to develop new diagnostic tool for early LD. In addition, the investigators will examine immune response in patients with various LD manifestations using flow cytometry, ELISA assay, and ELISpot assay. Finally, the investigators will perform whole genome sequencing of causative Bb-species isolated from patients to investigate potential differences in virulence and associations with clinical presentations.

Discussion:

This single-centre, observational cohort study will improve the understanding of immunological response in LD in children. It will also provide new information about the virulence of distinct LD causing Bb-genospecies and will test a new approach in the diagnosis of early LD.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting at the ED with differential diagnosis of LD according to the treating physician

Exclusion Criteria:

* Patients will be excluded in cases of primary or secondary immunodeficiency

Ages: 1 Month to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children from 0-17 years of age presenting with signs and symptoms suspicious for LD are included in the study. Previously healthy children with routine blood investigation are enrolled as healthy controls.
Sampling Method: Non-Probability Sample
Enrollment: 502 (Estimated)
Dates: Start 2024-04-02 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2028-11-01 (Estimated)

PRIMARY OUTCOMES:
Number of Bb-specific ASCs per 10^6 PBMCs | 10/2023 - 10/2026
  Method:
  Quantification of Bb-specific ASCs (IgM, IgG, IgA) per 10^6 PBMCs using ELISpot assay
  Time: 0 d (hospital admission), (1-14 d), 28 d, 3 m, and 6 m (after hospital admission)

SECONDARY OUTCOMES:
Measurement of percentage and median fluorescence intensity (MFI) of immune cell subsets in blood, CSF and SF | 10/2023 - 10/2028
  Method:
  Measuring percentage and MFI of innate and adaptive immune cell subsets using established panels for flow cytometry
  * innate immune cells: DC, GC, Nk-cells
  * adaptive immune cells: Tc-cells and Th-cell subsets (Th1, Th2, Th17, Treg), B-cells
  Time: 0 d (hospital admission), (1-14 d), 28 d, 3 m, and 6 m (after hospital admission)
Concentration of serum antibody levels (IU/mL) | 10/2023 - 10/2028
  Method:
  Measuring total serum IgM, IgG, IgA antibody levels using Enzyme-linked immunosorbant assay (ELISA)
  Time: 0 d (hospital admission), (1-14 d), 28 d, 3 m, and 6 m (after hospital admission)
Number of Bb-specific T cells per 10^6 PBMCs | 10/2023 - 10/2028
  Method:
  Quantification of Bb-specific INF-gamma-secreting T cells per 10^6 PBMCs using INF-gamma ELISpot assay.
  Time: 0 d (hospital admission), (1-14 d), 28 d, 3 m, and 6 m (after hospital admission)
Concentration of plasma and CSF cytokine/chemokine levels (pg/mL) | 10/2023 - 10/2028
  Method:
  Analysis of plasma and CSF cytokine/chemokine profiles using Multiplex Bead Array Kits
  * pro-inflammatory cytokines: interferon gamma (IFN-γ), Tumor necrosis factor A (TNF-α), IL-1, IL-17, IL-6 and IL-8
  * anti-inflammatory cytokines: IL-10 and IL-13
  * chemokines: Stromal cell-derived factor 1 (CXCL12), B cell-attracting chemokine 1 (CXCL13), IFN-γ inducible protein (IP-10/CXCL-10)
  Time: 0 d (hospital admission), (1-14 d), 28 d, 3 m, and 6 m (after hospital admission)
Portion of Bb positive LD patients by culture/PCR, identification of Bb species in LD patients | 10/2023 - 10/2028
  Method:
  Bb culture and PCR out of blood, CSF and SF samples
  Identification of Bb genospecies using PCR and whole genome sequencing (WGS)
  - Expected Bb genospecies: Bb sensu stricto, B. garinii, B. afzelii, B. spielmanii, B. mayonii
  Time: 0 d (hospital admission), (1-14 d), 28 d, 3 m, and 6 m (after hospital admission)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick M Meyer Sauteur, MD PhD, Principal Investigator — Division of infectious diseases Univesity Children's Hospital Zurich; Christoph Berger, MD, Study Director — Division of infectious diseases Univesity Children's Hospital Zurich
Locations (1):
- Chidren's Hospital Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Data will be handled with uttermost discretion and is only accessible to authorized personnel who require the data to fulfil their duties within the scope of the research. On the CRFs and other project specific documents, participants are only identified by a unique participant number. Biological material will be stored in coded manner with unique participant numbers in restricted areas at the Children's Research Center and the IMM. Collaborators will not be granted access to the key or any personal patient information.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Project data are stored for at least 15 years. Biological data will be collected for 5 years with a start in 2023 until 2028 and destroyed after 10 years of study closure.
Access Criteria: Access is authorized to personnel who require the data to fulfil their duties within the scope of the research.